CLINICAL TRIAL: NCT01498211
Title: Establishement of Normative Intra-epidermal Nerve Fiber Density Using Skin
Brief Title: Normative Data of Intra-epidermal Nerve Fiber Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4961
Record Dates: First submitted 2011-12-12; First posted 2011-12-23 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: volunteer
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biopsy (Experimental)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — 3 mm punch biopsy of the skin at the distal leg.

SUMMARY:
Intra-epidermal nerve fiber density can be assessed using skin biopsy. A decrease of this density is used to diagnose small fiber neuropathy, despite the absence of normative data in a selected normal population. To establish a normative set of data matched for age and sex is absolutely needed to evaluate the sensibility and specificity of this test.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 20-80 years old
* Normal subjects without pain and neurological impairment
* No history of neurological disorder
* Normal neurological examination
* Normal ECG
* Normal clotting sample from less than 6 months
* Available by phone

Exclusion criteria :

* History of alcoholic intoxication or chemotherapy
* History of diabetes, kidney insufficiency, monoclonal gammapathy, B/C hepatitis, HIV, coeliac disease, sicca syndrome, raynaud syndrome, systemic erythematous lupus, Fabry disease, amylosis, vascularitis
* Contraindication to xylocaïn with adrenalin
* At the site of biopsy : surgery, skin pathology, infection, vascular insufficiency
* Innate or acquired immunosuppression
* Innate or acquired clotting abnormality

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Measure density of intraepidermic nervous fibres by optical and electronic microscopy in a population of healthy witnesses according to the age and the sex. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas COLLONGUES, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (3):
- France (3):
  - CHU de Besançon, Besançon
  - CHU de Nancy, Nancy
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

REFERENCES:
- [Result] Collongues N, Samama B, Schmidt-Mutter C, Chamard-Witkowski L, Debouverie M, Chanson JB, Antal MC, Benardais K, de Seze J, Velten M, Boehm N. Quantitative and qualitative normative dataset for intraepidermal nerve fibers using skin biopsy. PLoS One. 2018 Jan 25;13(1):e0191614. doi: 10.1371/journal.pone.0191614. eCollection 2018. PMID 29370274